CLINICAL TRIAL: NCT06556862
Title: Exploration of Dalpiciclib Plus HDACi in HR+/HER2- Advanced Breast Cancer After Failure of CDK4/6 Inhibitor: a Phase II Study
Brief Title: Exploration of Dalpiciclib Plus HDACi in HR+/HER2- Advanced Breast Cancer After Failure of CDK4/6 Inhibitor
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Wang Tao, Professor, Beijing 302 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-211
Record Dates: First submitted 2024-08-05; First posted 2024-08-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: HR+/HER2- Advanced Breast Cancer
Keywords: post-CDK4/6 inhibitor; Dalpiciclib; HADCi; HR+/HER2- advanced breast cancer
MeSH Terms: interventions — dalpiciclib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib + plus HDACi (Experimental): Dalpiciclib + plus HDACi + Endocrine therapy (doctor's choice)
  Interventions: Drug: Dalpiciclib; Drug: Chidamide; Drug: Enitinostat

INTERVENTIONS:
Drug: Dalpiciclib — 100 mg/d, po., qd, administered on an empty stomach (fasting should be ensured at least 1 hour before and 1 hour after administration). The drug will be administered in a 28-day cycle, with continuously administration in the first 3 weeks (D1-21), and discontinuation in the fourth week (D22-28).
  Other Names: SHR6390
Drug: Chidamide — 25 mg/BIW, po. The interval between doses should not be less than 3 days (e.g. Monday and Thursday, Tuesday and Friday, Wednesday and Saturday, etc.), administered 30 minutes after meals
Drug: Enitinostat — 5mg/QW，po.

SUMMARY:
A phase II study to explore the efficacy and safety of dalpiciclib plus HDACi in HR+/HER2- advanced breast cancer after the failure of CDK4/6 inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study and sign the informed consent form
2. aged ≥ 18 years.
3. ECOG PS score: 0-2 points.
4. Expected survival ≥ 6 months.
5. Regionally recurrent or metastatic disease with histologically or cytologically confirmed ER+ and/or PR+ (≥ 10%), HER2- breast cancer that is not suitable for definitive excision or radiation therapy.
6. Previously received antitumor therapy: 1) previously received ≤1 line of chemotherapy for recurrent or metastatic breast cancer; 2) Disease recurrence and/or metastasis during or after treatment with Palbociclib or Abemaciclib or Ribociclib in the setting of (neo-)adjuvant therapy, or during treatment with palbociclib or Abemaciclib or Ribociclib in a metastatic setting or after disease progression; 3) No more than 3 lines of endocrine therapy have been previously received for recurrent or metastatic breast cancer. 4) Line number of previous chemotherapy ≤1 line
7. At least one extracranial measurable lesion as defined by RECIST v1.1;
8. The function of vital organs meets the requirements;

   * Absolute neutrophil count ≥ 1.5 × 10^9/L;
   * Platelets ≥ 90 × 10^9/L;
   * Hemoglobin ≥ 90g/L;
   * Total bilirubin (TBIL) ≤ 1.5 × ULN;
   * ALT and AST ≤ 2.5 × ULN;
   * Urea/blood urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN;
   * Left ventricular ejection fraction (LVEF) ≥ 50%;
   * The QT correction by the Fridericia formula (QTcF) is < 470 ms. INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN.
9. Subject recovers from any AE related to previous antitumor therapy before the first administration of the study drug (Grade ≤ 1)

Exclusion Criteria:

1. Previously received treatment with histone deacetylase inhibitor (HDACi);
2. Previously received Dalpiciclib;
3. MRI or lumbar puncture confirmed leptomeningeal metastasis;
4. Central nervous system metastasis is confirmed by imaging; The following conditions will be excluded: 1) asymptomatic brain metastases without immediate radiotherapy or surgery; 2) Previously received local treatment (radiotherapy or surgery) for brain metastases, stable for at least 4 weeks, and no symptomatic treatment (including glucocorticoids, mannitol, bevacizumab, etc.) for more than 2 weeks with clinical symptoms;
5. The participants presented with visceral crisis (such as lymphangitis carcinomatosis, bone marrow replacement, leptomeningeal metastasis, diffuse liver metastasis with abnormal liver function), rapid disease progression, and that is not suitable for endocrine therapy;
6. Participants had ascites, pleural effusion and pericardial effusion with clinical symptoms at baseline, which required drainage within 4 weeks before the first medication;
7. Inability to swallow, intestinal obstruction, or other factors that affect medication administration and absorption;
8. Subjects that are diagnosed with any other malignancy within 5 years prior to the study, excluding non-melanoma skin cancer treated with radical therapy, basal or squamous cell skin cancer or carcinoma in situ of the cervix and papillary thyroid.
9. The subject has undergone major surgery or major trauma or is expected to undergo major surgery within 4 weeks before the start of treatment;
10. A known history of allergy to the drug ingredient of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 Year
  Progression-free survival: The time to the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
ORR | 2 months
  Objective response rate
CBR | 2 Years
  Clinical benefit rate: CR+PR+SD≥6 months
DCR | 2 Years
  Disease Control Rate: CR+PR+SD
DoR | 2 Years
  The time from the beginning of CR or PR to the time when the tumor was first evaluated as PD or any cause of death.
OS | 2 Years
  The time from the beginning of treatment to the time of death caused by any cause
Safety | AE recorded from infromed consent to 28 days after treatment completion
  Adverse events (AE), serious adverse events (SAE), and immune-related adverse events (irAE), in accordance with the NCI-CTC AE version 5.0 criteria. AE recorded from infromed consent to 28 days after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China